CLINICAL TRIAL: NCT02732951
Title: A Randomized, Double-masked, Placebo-controlled Exploratory Study to Evaluate Pharmacodynamics, Safety and Tolerability of Orally Administered BI 1026706 for 12 Weeks in Patients With Mild Visual Impairment Due to Center-involved Diabetic Macular Edema (DME)
Brief Title: Safety and Effect on Central Retinal Thickness of BI 1026706 in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1320.22; 2015-003529-33 (EudraCT Number)
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- BI 1026706 (Experimental)
  Interventions: Drug: BI 1026706
- Placebo (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1026706
  Arms: BI 1026706
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a proof of mechanism trial to explore the effect of BI 1026706 on the central retinal thickness and to evaluate safety and tolerability of BI 1026706 administered orally for 12 weeks in patients with mild vision impairment due to center-involved DME

ELIGIBILITY:
Inclusion criteria:

* Patients 18 years of age and older
* Male patients or female patients of non-childbearing potential
* Diagnosis of Diabetes mellitus type 1 or type 2
* Retinal thickening due to Diabetic macular edema (DME) involving the center of the macula in the study eye as confirmed by the Investigator on clinical exam
* Center-involved DME confirmed on Spectral-Domain Optical Coherence Tomography (SD-OCT) with central subfield thickness (CSFT) of at least 300 µm in the study eye at screening, confirmed by Central Reading Centre
* Best corrected visual acuity ETDRS (Early Treatment Diabetic Retinopathy Study) letter score in the study eye of 84 or below, but at least 70 at screening
* Further inclusion criteria apply

Exclusion criteria:

* Macular edema considered to be due to other causes than DME in the study eye
* Additional eye disease in the study eye that, in the opinion of the Investigator, might affect macular edema or could compromise or alter visual acuity during the course of the trial
* Anterior segment and vitreous abnormalities in the study eye that would compromise the adequate assessment of the best corrected visual acuity or an adequate examination of the posterior pole
* Intraocular surgery in the study eye within 4 months prior to randomization or planned intraocular surgery, including cataract, during the study period
* Proliferative diabetic retinopathy or iris neovascularisation in the study eye
* Aphakia in the study eye
* Any indication that requires immediate treatment or for which treatment is expected in the study eye with anti-Vascular Endothelial Growth Factor (VEGF) or with laser photocoagulation during the period, as per Investigator's judgment
* History of prior laser photocoagulation or other surgical, intravitreal or peribulbar treatment in the study eye within 4 months prior to randomization, either for DME or an ocular condition other than DME
* History of fluocinolone acetonide intravitreal implant in the study eye
* Application of intraocular corticosteroids in the study eye within 2 years prior to randomization in phakic eyes or 9 months in pseudophakic eyes
* History of topical steroid or nonsteroidal anti-inflammatory drugs (NSAID) treatment in the study eye within 30 days prior to randomization
* Systemic anti-VEGF or pro-VEGF treatment within 4 months prior to randomization
* Initiation of intensive insulin treatment (multiple daily injections or a pump) within 3 months prior to randomization or plans to do so in the next 4 months
* Change in oral antidiabetic medication within 3 months prior to randomization
* Patients with a clinically relevant abnormal screening haematology, blood chemistry, or urinalysis
* Renal impairment with estimated creatinine clearance < 30 mL/min (as calculated by Cockcroft-Gault equation)
* Myocardial infarction or unstable angina pectoris within 3 months before randomization
* Uncontrolled arterial hypertension defined as a single measurement of systolic >180 mmHg, two consecutive measurements of systolic >160 mmHg, or diastolic >100mmHg on optimal medical regimen
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (35):
- Belgium (2):
  - Brussels-UNIV Brugmann -Horta, Brussels
  - Leuven - UNIV UZ Leuven (Sint-Rafaël), Leuven
- France (5):
  - HOP Nord, Marseille
  - HOP Hôtel-Dieu, Nantes
  - HOP Lariboisière, Paris
  - Hosp National 15-20, Ophtalmo, Paris, Paris
  - HOP Pierre Paul Riquet, Toulouse
- Germany (8):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Augen Zentrum Nordwest, Ahaus, Ahaus
  - Kamppeter Augenzentrum, Bayreuth, Bayreuth
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Augenarzt Dr. Dunker und Kollegen, Troisdorf, Troisdorf-Sieglar
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Greece (3):
  - Attikon, Panepistimiako Geniko Nosokomeio, Athens
  - University General Hospital of Heraklion, Herakleion,Crete
  - University of Patras Medical School, Pátrai
- Hungary (3):
  - Uzsoki Street Hospital, Budapest, Budapest
  - BAZ County Hospital, Ophtalmology Department, Miskolc, Miskolc
  - Univ.Szeged;Szent-Gyorgyi;Albert Heal.Cent.Ophtalmology Dep, Szeged
- Portugal (4):
  - Hospital de Braga-Escala Braga, Braga
  - AIBILI - Association for Innovation and Biomedical Research on Light and Image, Coimbra
  - Centro Hospitalar São João,EPE, Porto
  - Hospital de Vila Franca de Xira, Vila Franca de Xira
- Spain (5):
  - Hospital Dos de Maig, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital La Paz, Madrid
  - Instituto Oftalmológico Gómez-Ulla, Santiago de Compostela
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (5):
  - Frimley Park Hospital, Frimley
  - Royal Surrey County Hospital, Guildford
  - Moorfields Eye Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Southampton General Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was randomised, double-blind, placebo-controlled, parallel-group trial to evaluate pharmacodynamics, safety and tolerability of orally administered Boehringer Ingelheim (BI) 1026706 for 12 weeks in patients with Diabetic Macular Oedema (DME).
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites which would then ensure that all patients met all inclusion/exclusion criteria. Patients were not to be randomized to trial treatment if any one of the specific entry criteria were violated.
Groups:
- Placebo Matching to BI 1026706: Patients were administered film-coated tablet of placebo to match 100 mg BI 1026706 twice daily orally for 12 weeks.
- BI 1026706: Patients were administered film-coated tablet of 100 mg BI 1026706 twice daily orally for 12 weeks.
Period: Overall Study
Arm/Group | Placebo Matching to BI 1026706 | BI 1026706
Started (Randomised and treated) | 53 | 52
Completed (Completed trial) | 48 | 46
Not Completed | 5 | 6
Not completed — Other than listed | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 4 | 4
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS includes all patients who were treated with at least 1 dose of trial drug, either BI 1026706 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching to BI 1026706 | BI 1026706 | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: TS
  Years | 62.2 (9.7) | 63.9 (8.7) | 63.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 14 | 14 | 28
    Male | 39 | 38 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    Hispanic or Latino | 4 | 4 | 8
    Not Hispanic or Latino | 35 | 43 | 78
    Unknown or Not Reported | 14 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: TS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 38 | 47 | 85
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 14 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Subfield Foveal Thickness (CSFT) at Week 12
Description: The change from baseline in CSFT at Week 12 and the BI 1026706 effect was compared between the BI 1026706 treatment group and the placebo group as measured by Spectral-domain Optical Coherence Tomography (SD-OCT). Baseline was defined as the CSFT value measured at the visit when patients were randomised. Mean presented here is an adjusted mean.
Time Frame: Baseline and Week 12
Population: Full analysis set (FAS): FAS includes all patients who were randomised, treated with at least 1 dose of BI 1026706 or placebo, and with a baseline and at least one post randomisation central subfield foveal thickness (CSFT) measurement.
Measure: Mean (Standard Deviation); unit: Micrometre [μm]
Arm/Group | Placebo Matching to BI 1026706 | BI 1026706
Number analyzed (Participants) | 47 | 47
Micrometre [μm] | -6.19 (11.61) | 10.26 (11.64)
Statistical Analysis 1: Comparison: Placebo Matching to BI 1026706 vs BI 1026706; Null hypothesis = The CSFT change from baseline at Week 12 is equal in both groups; Test type: Other; p = 0.3199, Mixed model for repeated measurements; Kenward-Roger approximation was used for denominator degrees of freedom; Adjusted Mean = 16.45, 95% CI 2-sided [-16.23 to 49.13], Standard Error of Mean 16.45 — Fixed effects of treatment, prior anti-diabetic macular oedema treatment status, visit, treatment by visit interaction, baseline, baseline by visit interaction; patient as a random effect; unstructured covariance matrix for within patient errors

2. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs), Investigator Defined Drug-related Adverse Events (AEs) and Adverse Events of Special Interest (AESIs)
Description: Number of subjects with serious adverse events (SAEs), Investigator defined drug-related Adverse events (AEs) and adverse events of special interest (AESIs) comparing the BI 1026706 treatment group with the placebo group is presented.
Time Frame: From first drug administration until 4 days after last drug administration, up to 89 days.
Population: as for baseline characteristics
Measure: Number; unit: Count of participants
Arm/Group | Placebo Matching to BI 1026706 | BI 1026706
Number analyzed (Participants) | 53 | 52
Count of participants
  Total with SAEs | 2 | 7
  Investigator defined drug-related AE | 7 | 7
  AESIs | 0 | 1

ADVERSE EVENTS:
Time Frame: From first drug administration until 4 days after last drug administration, up to 89 days.
Arm/Group | Placebo Matching to BI 1026706 | BI 1026706
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/53 | 7/52
Other Adverse Events (participants affected / at risk) | 12/53 | 14/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching to BI 1026706 (N=53) | BI 1026706 (N=52)
Myocardial infarction (Cardiac disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1
Reactive perforating collagenosis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching to BI 1026706 (N=53) | BI 1026706 (N=52)
Visual acuity reduced (Eye disorders) | 2 | 3
Nasopharyngitis (Infections and infestations) | 4 | 6
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Headache (Nervous system disorders) | 1 | 4
Somnolence (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT02732951/SAP_000.pdf
  • Study Protocol (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT02732951/Prot_001.pdf